CLINICAL TRIAL: NCT06824064
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study of RBS2418 Plus Best Supportive Care (BSC) in Subjects With Advanced, Metastatic, and Progressive Colorectal Cancer
Brief Title: Evaluation of RBS2418 in Patients With Advanced, Metastatic, and Progressive Colorectal Cancer
Acronym: VISTA-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Riboscience, LLC. (Industry)
Collaborators: Tam Anh Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBS2418-2001
Record Dates: First submitted 2025-01-30; First posted 2025-02-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer; Advanced Colorectal Cancer
Keywords: Advanced, Metastatic, Progressive Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: EG+ [ENPP1 and cGAS(Cyclic GMP-AMP synthase) positive] RBS2418 plus Best Supportive Care (Active Comparator): RBS2418: 200 mg (2 RBS2418 capsules), PO (by mouth), BID (twice a day) plus Best Supportive Care
  Interventions: Drug: RBS2418
- Group B: EG+ (ENPP1 and cGAS positive) Placebo plus Best Supportive Care (Placebo Comparator): Placebo: 2 placebo capsules, PO, BID plus Best Supportive Care
  Interventions: Drug: Placebo
- Group C: EG- (ENPP1 and/or cGAS negative) RBS2418 plus Best Supportive Care (Active Comparator): RBS2418: 200 mg (2 RBS2418 capsules), PO, BID plus Best Supportive Care
  Interventions: Drug: RBS2418
- Group D: EG- (ENPP1 and/or cGAS negative) Placebo plus Best Supportive Care (Placebo Comparator): Placebo: 2 placebo capsules, PO, BID plus Best Supportive Care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBS2418 — RBS2418 is a specific immune modulator that works through the inhibition of ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) and is designed to lead to anti-tumor immunity by protecting endogenous 2'-3'-cyclic guanosine monophosphate-adenosine monophosphate (cGAMP) from hydrolysis and leading to the activation of antigen-presenting cells followed by T cell activation.
  Arms: Group A: EG+ [ENPP1 and cGAS(Cyclic GMP-AMP synthase) positive] RBS2418 plus Best Supportive Care; Group C: EG- (ENPP1 and/or cGAS negative) RBS2418 plus Best Supportive Care
Drug: Placebo — Placebo to Match RBS2418
  Arms: Group B: EG+ (ENPP1 and cGAS positive) Placebo plus Best Supportive Care; Group D: EG- (ENPP1 and/or cGAS negative) Placebo plus Best Supportive Care

SUMMARY:
RBS2418 is a specific immune modulator that works through the inhibition of ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) and is designed to lead to anti-tumor immunity by protecting endogenous 2'-3'-cyclic guanosine monophosphate-adenosine monophosphate (cGAMP) from hydrolysis and leading to the activation of antigen-presenting cells followed by T cell activation. The hypothesis is that RBS2418 versus placebo will be generally safe, well-tolerated, immunogenic, and will lead to anti-tumor responses in adult subjects for the treatment of advanced, metastatic, and progressive colorectal cancer (CRC).

DETAILED DESCRIPTION:
In this Phase 2a study, subjects must have failed, been unable to tolerate, or declined to take known standard-of-care (SOC) therapies. Subjects must have measurable disease per RECIST 1.1, an Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1 or 2, and predicted life expectancy of greater or equal to 3 months.

Up to approximately 150 subjects will be enrolled and will receive therapy as part of their respective treatment group. Subjects will receive study treatment of RBS2418 or Placebo to Match plus Best Supportive Care with a treatment period consisting of 21-day cycles up to two years or until there is progressive disease (PD), death, withdrawal, or study completion, whichever comes first.

Adverse events (AEs) will be monitored throughout the study and graded in severity according to the guidelines outlined in the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. AEs will be collected until up to 30 days after the end of treatment or until resolution, whichever comes first. Serious Adverse Events (SAEs) will be collected for 90 days after the end of treatment, or if the subject initiates new anti-cancer therapy, then 30 days after the end of treatment, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age on the day of signing informed consent.
2. Male and female subjects with advanced, metastatic, progressive CRC who have received, been ineligible for, intolerant to, or declined all approved standard of care (SOC) therapies for metastatic CRC, as per local SOC treatment regimens. Additionally, subjects must have documented PD based on two scans performed within 2 to 4 months of study initiation.
3. Have histologically or cytologically confirmed CRC diagnosis based on pathology report.
4. Willing to submit a pre-treatment tissue sample (archival, or fresh tissue if archival is not available).

Exclusion Criteria:

1. Any approved anti-cancer therapy including chemotherapy, targeted small molecule therapy, systemic immunotherapy, or radiation therapy within 2 weeks prior to the first dose of study treatment; or if subject has not recovered (i.e., ≤ to Grade 1 or returned to baseline level) from AEs due to a previously administered agent; the following exceptions are allowed:

   * Palliative radiotherapy for bone metastases or soft tissue lesions should be completed >7 days prior to the first dose of study treatment.
   * Hormone-replacement therapy or oral contraceptives.
   * Subjects with Grade 2 neuropathy or Grade 2 alopecia.
2. Subjects with evidence of rapid progression on prior therapy resulting in rapid clinical deterioration.
3. Malignancies other than indications open for enrollment within 3 years prior to Day 1, except for those with negligible risk of metastasis or death treated with expected curative outcome, undergoing active surveillance, or treatment-naïve for indolent tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From randomization until the first radiographic documentation of objective progression or death from any cause, assessed up to 2 years.
  Time in months from randomization until the first radiographic documentation of objective progression, as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, or death from any cause
Overall Survival | From randomization until death from any cause, assessed up to 2 years.
  Time in months from the date of randomization to the date of death from any cause

SECONDARY OUTCOMES:
Duration of Response (DOR) | From initial response to disease progression or death, assessed up to 2 years.
  DOR is defined as the time in months from initial response [when complete response (CR) or partial response (PR) is first determined] to disease progression or death, whichever comes first.
Disease Control Rate (DCR) | From randomization to end of treatment or disease progression, assessed up to 2 years.
  DCR is defined as the percentage of subjects who achieve a complete response (CR), a partial response (PR) or stable disease (SD).

CONTACTS AND LOCATIONS:
Locations (3):
- Community Clinical Trials, Kingwood, Texas, United States
- Vietnam (2):
  - Tam Anh TP. Ho Chi Minh General Hospital, Ho Chi Minh City, Ho Chi Minh City
  - Tam Anh, Ha Noi General Hospital, Hà Nội

IPD SHARING:
Plan to Share IPD: No